CLINICAL TRIAL: NCT05835557
Title: Physiological Outcomes of High-intensity Interval Training With Post-exercise Blood Flow
Brief Title: Physiological Outcomes of High-intensity Interval Training With Post-exercise Blood Flow Restriction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanyang Technological University (Other)
Responsible Party: Principal Investigator, Stephen Burns, Associate Professor, Nanyang Technological University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IRB-2023-235
Record Dates: First submitted 2023-04-05; First posted 2023-04-28 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Exercise Performance

STUDY DESIGN:
Intervention Model Description: Two groups exposed to 9 sessions of high intensity short interval training with or without blood flow restriction between sets of exercise.
Who Masked: Participant
Masking Description: Sham treatment of altitude exposure in an environmental chamber.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Blood flow restriction with short interval training (BFR-ST) (Experimental): 9 sessions of high intensity short interval training with blood flow restriction.
  Interventions: Other: BFR-ST
- Sham altitude with short interval training (ST) (Sham Comparator): 9 sessions of high intensity short interval training in an altitude chamber.
  Interventions: Other: ST

INTERVENTIONS:
Other: BFR-ST — Undergo 9 sessions of high intensity short interval training involving 3 sets of 8-10 repetitions of 30 secs interval cycling and 30 secs recovery at 100-110% of maximal aerobic power. In between sets there will be 3 mins of passive rest. Blood flow restriction will be applied for 2 mins during the passive rest at 80% of limb occlusion pressure.
  Arms: Blood flow restriction with short interval training (BFR-ST)
Other: ST — Undergo 9 sessions of high intensity short interval training involving 3 sets of 8-10 repetitions of 30 secs interval cycling and 30 secs recovery at 100-110% of maximal aerobic power. In between sets there will be 3 mins of passive rest. Cycling will be conducted in an environmental chamber and participants informed that the altitude is set to 2500m - actual altitude will be sea level.
  Arms: Sham altitude with short interval training (ST)

SUMMARY:
This research study revolves around the physiological outcomes of using post-exercise blood flow restriction (BFR) with high intensity short interval training (ST) The main aims of this study are to compare (i) aerobic performance outcomes, and (ii) anaerobic and muscular performance outcomes - between 2 groups of participants after either undergoing 3 weeks of ST + post-exercise BFR (BFR-ST) or traditional ST.

DETAILED DESCRIPTION:
This research study revolves around the physiological outcomes of using post-exercise blood flow restriction (BFR) with high-intensity interval exercise training (HIIT), specifically high intensity short interval training (ST) protocol of 30s work, 30s rest, for the recreational endurance athlete. In previous research, it has been shown that using BFR during rest intervals of a ST protocol would elicit greater physiological stresses in terms of higher heart rate, greater muscle activation, reduced oxygenation within the muscle tissue during exercise, and increased blood lactate post-exercise as compared with the control condition. However, the physiological outcomes of this type of training method over a longer-term (9 sessions over 3 weeks) have not been explored. The main aims of this study is to compare the physiological outcomes, - (i) aerobic performance outcomes, and (ii) anaerobic and muscular performance outcomes - between 2 groups of participants after either undergoing 3 weeks of ST + post-exercise BFR (BFR-ST) or traditional ST . The hypotheses for this study are: the BFR-ST group would experience a (i) greater improvement in maximal aerobic capacity, function and time trial performance and, (ii) greater improvement in anaerobic power and capacity as well as muscular strength and power, as compared with the ST group.

ELIGIBILITY:
Inclusion Criteria:

* Male
* 18-40 years
* Actively performing endurance exercise (running or cycling) for at least 2 sessions (1 - 1.5h) per week
* Healthy (free from illnesses) and no musculoskeletal injuries for the past 6 months
* No history of cardiometabolic, vascular diseases or similar conditions (e.g., high blood pressure, peripheral vascular diseases, heart diseases, metabolic syndrome, diabetes, stroke, etc.).
* Pass the pre-participation health screening tests - Physical Activity Readiness Questionnaire for Everyone (PAR-Q+) and Australian Institute of Sport Blood Flow Restriction (AIS BFR) pre-screening questionnaire (no history of any risk factors).
* Achieve a maximum oxygen uptake (VO2max) of ≥40ml/kg/min during a maximal aerobic power cycling screening test.
* Non-smoker
* Drink alcohol less than 3 times each week and less than 3 drinks each time

Exclusion Criteria:

* Persons with any form of illnesses and/or musculoskeletal injuries for the past 6 months
* Any history of cardiometabolic, vascular diseases or similar conditions which may worsen with the use of blood flow restriction during exercise
* Fail the pre-participation health screening tests
* Below 40ml/kg/min VO2max during maximal aerobic power cycling test
* Smoker
* Consumption of alcohol beyond that stated in the inclusion criteria.
* History of asthma or taking medication for asthma.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Males
Enrollment: 40 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Maximum oxygen uptake and power | Will be assessed at baseline (Day 0 - Pre) and the change in this outcome 24 hours after 9 sessions of training over 3 weeks (Post)
20 km Cycling time trial | Will be assessed at baseline (Day 0 - Pre) and the change in this outcome 24 hours after 9 sessions of training over 3 weeks (Post)
Wingate test of anaerobic power | Will be assessed at baseline (Day 0 - Pre) and the change in this outcome 24 hours after 9 sessions of training over 3 weeks (Post)
  Peak and mean power and rate of fatigue

SECONDARY OUTCOMES:
Exercise economy | Will be assessed at baseline (Day 0 - Pre) and the change in this outcome 24 hours after 9 sessions of training over 3 weeks (Post)
  Oxygen uptake at a fixed load of 50% of maximum aerobic power
Isometric mid-thigh pull | Will be assessed at baseline (Day 0 - Pre) and the change in this outcome 24 hours after 9 sessions of training over 3 weeks (Post)
  Maximal strength assessment of lower body
Countermovement jump height | Will be assessed at baseline (Day 0 - Pre) and the change in this outcome 24 hours after 9 sessions of training over 3 weeks (Post)
  Vertical jump height assessment

CONTACTS AND LOCATIONS:
Locations (1):
- Human Bioenergetics Laboratory, National Institute of Education, Nanyang Technological University, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Yes
All published data will be placed into the Data Repository of Nanyang Technological University National Institute of Education for public access upon publication.
Supporting Information: Analytic Code
Time Frame: Upon publication - permanent repository
Access Criteria: Public repository - exact web address available upon publication.
URL: http://researchdata.nie.edu.sg/

REFERENCES:
- [Derived] Chua MT, Sim A, Aziz AR, Polglaze T, Burns SF. Blood Flow Restriction during Rest Periods of High-Intensity Interval Training Enhances Endurance Performance: A Randomized Placebo-Controlled Study. Med Sci Sports Exerc. 2026 Jan 1;58(1):86-98. doi: 10.1249/MSS.0000000000003834. Epub 2025 Aug 12. PMID 40792614